CLINICAL TRIAL: NCT06150820
Title: A Study to Evaluate Seroprevalence of Antibodies to AAV8 and Assessment of Biomarkers in Patients With Late-Onset Pompe Disease
Brief Title: A Study About Antibody Levels and Biomarkers in the Blood in People With Late-onset Pompe Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AT845-02
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pompe Disease (Late-onset)
Keywords: Pompe Disease (Late-onset); Antibodies to AAV8; Biomarkers
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Late-Onset Pompe Disease (Other): Adolescent or adult participants with LOPD.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No investigational drug will be administered to participants in this study.

SUMMARY:
Pompe disease is a genetic condition which causes muscle weakness over time. People with Pompe disease have a faulty gene that makes an enzyme called acid alpha-glucosidase (or GAA). This enzyme breaks down a type of sugar called glycogen. Without this enzyme, there is a build-up of glycogen in the cells of the body. This causes muscle weakness and other symptoms. Pompe disease can happen at any age, but in late-onset Pompe disease, symptoms generally start from 12 months old onwards.

The standard treatment for people with Pompe disease is to receive regular infusions of the GAA enzyme. This is known as enzyme replacement therapy. However, people can build up antibodies against the GAA enzyme over time.

Gene therapy is used to treat conditions caused by a faulty gene. It works by replacing the faulty gene with a working gene inside the cells of the body. The working gene is delivered into the cells using certain viruses as carriers (vectors). Viruses are often used as carriers as they can easily get inside cells. The genetic material of the original virus is replaced with the working gene, so only the working gene gets inside the cells. A common virus used as a carrier in gene therapy is the adeno-associated virus (or AAV). This is like an adenovirus, which causes the common cold.

The original type of AAV does not cause any harm to humans. However, people that have previously been infected with the original type of AAV may have built up antibodies against AAV. These antibodies may stop the AAV carrier with the working gene getting inside the cells.

Researchers want to learn more about antibody levels against AAV and the GAA enzyme in people with late-onset Pompe disease. They also want to learn about other substances in the blood that provide more information about late-onset Pompe disease. These are known as biomarkers.

In this study, older teenagers and adults with late-onset Pompe disease will take part. They will not have had gene therapy using AAV. There will be 2 groups - those who have never had enzyme replacement therapy, and those who have had enzyme replacement therapy for 6 months or more. No study treatment will be given during the study, but blood and urine samples will be taken for testing.

The main aims of the study are to check antibody levels against AAV8 (a type of AAV) in people with late-onset Pompe disease who had not received any treatment using AAV, to check antibody levels against the GAA enzyme in people previously treated with GAA as part of enzyme replacement therapy, to check levels of biomarkers for Pompe disease, and to check for medical problems.

In the study, people will visit the study clinic several times. Some visits may be in the person's home. The first visit is to check if they can take part. Those who can take part will have a medical examination, and have their vital signs checked. Vital signs include blood pressure, heart rate, breathing rate and temperature. Blood samples will be taken to check antibody levels against the GAA enzyme and against AAV8. Blood and urine samples will also be taken to check for biomarkers for Pompe disease. Blood and urine samples will be taken about every 4 months for up to 2 years.

DETAILED DESCRIPTION:
No investigational drug will be administered to participants in this study. Blood and urine will be collected as part of the study. The duration of the study is approximately 2 years, participants may withdraw at any time.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a documented clinical diagnosis of LOPD.
* Participant is enzyme replacement therapy ERT-naïve (ERT-N) or if the participant is currently taking an approved ERT treatment or is participating in an ERT-interventional study, the ERT must have been received for at least 6 months or more (ERT-experienced [ERT-E]).
* Participant is willing and able to comply with study visits and procedures.
* Participant agrees to not start participating in any other clinical study involving an investigational study treatment, including ERT, while participating in this study.

Exclusion Criteria:

* Participant previously received an AAV-related product (any serotype).
* Participant is currently participating in a Pompe-related interventional study (other than ERT-interventional studies) or has received gene or cell therapy.
* Participant requires any invasive or noninvasive ventilation support while awake and upright (non-invasive support while sleeping with either continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) is acceptable for eligibility).
* Participant is unable to ambulate (assistive devices [e.g., cane or walker] are acceptable for eligibility).
* Participants who have received any ERT for less than 6 months as of the Baseline visit are not eligible.

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of total antibodies to AAV8 | Up to 2 years
  Antibodies to AAV8 will be recorded from serum blood samples collected.
Occurrence of neutralizing antibodies to AAV8 | Up to 2 years
  Antibodies to AAV8 will be recorded from serum blood samples collected.

SECONDARY OUTCOMES:
Seroconversion of antibodies to AAV8 over time | Up to 2 years
  Seroconversion of antibodies to AAV8 will be recorded from serum blood samples collected.
Creatine kinase [CK] levels | Up to 2 years
  CK levels will be recorded from blood plasma samples collected.
Urine glucose tetrasaccharide [Glc4]/hexose tetrasaccharide [Hex4] over time | Up to 2 years
  Glc4/Hex4 will be recorded from urine samples collected.
Occurrence of anti-GAA antibodies in participants on ERT | Up to 2 years
  Anti-GAA antibodies will be recorded from serum blood samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Gene Therapies
Locations (53):
- United States (10):
  - Emory Clinic, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of UTAH - PPDS, Salt Lake City, Utah
  - Lysosomal and Rare Diseases Research and Treatment Center, Inc., Fairfax, Virginia
- Australia (2):
  - AU61003, Adelaide
  - AU61001, Herston
- Brazil (3):
  - BR55003, Flamengo
  - BR55002, Porto Alegre
  - BR55001, São Paulo
- Canada (2):
  - CN15003, Edmonton
  - CA15001, Montreal
- France (8):
  - FR33006, Angers
  - FR33009, Garches
  - FR33005, Lille
  - FR33007, Limoges
  - FR33002, Marseille
  - FR33003, Nantes
  - FR33004, Nice
  - FR33001, Strasbourg
- Germany (4):
  - DT49005, Bonn
  - DT49004, Essen
  - DT49003, Höchheim
  - DT49006, Münster
- Italy (9):
  - IT39002, Florence
  - IT39005, Gussago
  - IT39012, Messina
  - IT39009, Milan
  - IT39011, Milan
  - IT39008, Pavia
  - IT39006, Pisa
  - IT39004, Roma
  - IT39003, Udine
- Japan (2):
  - National Center of Neurology and Psychiatry, Kodaira-Shi
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku
- Spain (7):
  - ES34003, Albacete
  - ES34004, Barcelona
  - ES34009, Donostia / San Sebastian
  - ES34007, L'Hospitalet de Llobregat
  - ES34001, Madrid
  - ES34005, Madrid
  - ES34002, Valencia
- Taiwan (3):
  - TW88601, Taipei
  - TW88602, Taipei
  - TW88603, Taoyuan
- United Kingdom (3):
  - UK44003, Cambridge
  - UK44001, Newcastle upon Tyne
  - UK44004, Salford

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.